CLINICAL TRIAL: NCT01021787
Title: Dermal Penetration of the Titanium Dioxide in Anthelios SX SPF 40 Sunscreen Cream With Micronized TiO2 and Anthelios SX SPF 40 Cream (With Pigmentary TiO2) Into the Stratum Corneum of Compromised (Induced Sunburn) Human Skin
Brief Title: Dermal Penetration of the Titanium Dioxide in Anthelios SX SPF40 Cream
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Loreal USA (Industry)
Responsible Party: Jean Grieve, Assistant Vice President, L'Oreal USA Products Inc.
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: PEN.750.06
Record Dates: First submitted 2009-11-25; First posted 2009-11-30 (Estimated); Last update posted 2011-06-14 (Estimated); Status verified 2009-11

CONDITIONS: Sunburn
Keywords: Sun Protection
MeSH Terms: conditions — Sunburn | interventions — titanium dioxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Titanium dioxide — Topical cream

SUMMARY:
To determine the penetration of micronized and pigmentary TiO2 in Formulas 283419 2 and 760.001 into the stratum corneum of Compromised (Induced Sunburn) human skin via skin stripping of human subjects.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must:

  1. be between the ages of 18 and 65.
  2. agree to not participate in any other product evaluations or clinical evaluations during the course of this study.
  3. have read, understood and signed an Informed Consent Form.
  4. have intact skin in the treatment area.
  5. have fair skin - Skin Types I, or II - as defined in Appendix II.
  6. be able to understand and willing to follow all study procedures and restrictions.

Exclusion Criteria:

Subjects will be excluded from participating in the study if they:

1. are female and are pregnant or lactating [must be using an acceptable method of birth control if of child bearing potential].*
2. exhibit any visible symptoms of skin disease, such as psoriasis or eczema, or skin abnormality (including active dermal lesions, uneven skin tone or scars) which might interfere with interpretation of the study results. The presence of nevi, blemishes, or moles will be acceptable if, in the Investigator's judgement, they will not interfere with the study results or skin stripping procedures.
3. have a history of allergic responses to sunscreens or other products similar to those included in this study.
4. have very dry or scaly skin on the test site.
5. have diabetes.
6. have a history of abnormal responses to sunlight, such as a phototoxic or photoallergic response.
7. have an existing sunburn or suntan, or been to a tanning booth which would interfere with interpretation of the study results.
8. have used self tanners within the past two weeks.
9. have excessive hair at the test site area which could, in the opinion of the investigator, interfere with the interpretation of the results.
10. have participated in a research drug trial or patch test within six weeks of beginning this study.
11. have a known sensitivity to Scotch 600 Transparent Tape.
12. are currently receiving, or within the past two weeks received, topical or systemic medication which could, in the opinion of the investigator, interfere with the interpretation of the results, affect the safety of the subject, or which may change the body's response to ultraviolet light.
13. are currently taking any of the drugs listed on the next page. In addition, the use of St. John's Wort or other similar dietary supplements, aspirin or OTC ibuprofen is contraindicated for the duration of the study. Low dose daily aspirin use, 81 mgs, taken for heart attack prevention is excluded.

    * Acceptable methods of birth control that can be used during the course of the study are: oral contraceptive pill, intrauterine device, patch, injection, condom with spermicide, partner vasectomy, bilateral tubal ligation, abstinence or evidence of non childbearing potential (i.e., post-menopausal [one year without menstrual period], hysterectomy or bilateral ovariectomy).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Determine degree of penetration of TiO2 down to 16 -20 tape strips of human skin | Single application

CONTACTS AND LOCATIONS:
Locations (1):
- Hill Top Research, Winnipeg, Manitoba, Canada